CLINICAL TRIAL: NCT03656887
Title: Screening for Hypoglycemia in an Institutionalized Elderly Diabetic Population.
Acronym: HAGED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOUILLET 2018
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Old Age; Institutionalized in EHPAD (French Nursing Home); Diabetes; Hypoglycemic Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous interstitial glucose sensor — Installing and removing the sensor
Other: Sensor Scan — Scan of the sensor, using the Freestyle Pro free version reader, at installation then before removal after 14 days.

SUMMARY:
Diabetes is a major public health problem that has been growing steadily in recent years. Its prevalence is very high in the elderly, in whom there is an increased risk of hypoglycemia.

Hypoglycaemia in elderly diabetics has serious consequences:

* increased mortality,
* increased cardiovascular morbidity,
* increased risk of falling,
* impairment of quality of life.
* Hypoglycaemia is also a risk factor for dementia in type 2 diabetes. The frequency of asymptomatic and atypical hypoglycemia has been shown to be greater in the elderly, but the exact prevalence of hypoglycemia in the elderly remains unknown.

Elderly diabetic patients in institutions are particularly fragile and have more frequent cognitive problems than non-diabetic subjects. A study conducted in this population of patients showed that a third of them had HbA1C <6.5%, which suggests a higher frequency of hypoglycemia though the figures were not available.

We therefore decided to conduct a study to assess the frequency of hypoglycemia in order to better understand the contributing factors and to improve the management of this fragile population.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* diabetic patient receiving treatment which could result in hypoglycemia: insulin and/or sulfonamide and/or glinides
* institutionalized patient in an EHPAD
* patient over 60 years of age

Exclusion Criteria:

- person not affiliated to a national health insurance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient institutionalized in EHPAD
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic events (<70 mg/dl) demonstrated by continuous interstitial glucose monitoring over the study period. | Day 14
Number of hypoglycemic events (<70 mg/dl) detected by capillary blood glucose measurement or clinical signs suggestive of hypoglycemia. | Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Bouillet B, Tscherter P, Vaillard L, Nonciaux C, Hourdain P, Ravier A, Rouland A, Petit JM, Verges B, Quilot E. Frequent and severe hypoglycaemia detected with continuous glucose monitoring in older institutionalised patients with diabetes. Age Ageing. 2021 Nov 10;50(6):2088-2093. doi: 10.1093/ageing/afab128. PMID 34324624